CLINICAL TRIAL: NCT04371328
Title: Emergency Management in a Dedicated Respiratory Unit of Patients With a Possible COVID-19 Infection (Unit "COVID Possible")
Brief Title: Emergency Management in a Dedicated Respiratory Unit of Patients With a Possible COVID-19 Infection
Acronym: RECOP
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0094
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Emergencies
Keywords: COVID 19; aspecific respiratory symptomatology
MeSH Terms: conditions — Emergencies; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: RECOP unit patient — All patients admit in RECOP unit for dyspnea can be included in this study if patient is agree. Then, doctor collects demographic variables, the usual history and treatments, the characteristics of the episode (symptomatology, evolution, treatment taken) and the data from the initial clinical examination will be identified.
  30 days after inclusion, virological status and mortality will be collect

SUMMARY:
This research aims to improve knowledge of the epidemiology of patients consulting in the COvid Possible REspiratory Units (RECOP unit). Indeed, the epidemic linked to COVID19 affects France and impacts its health system. The reception of all intermediate patients will be on the Emergency Structures (SU). Indeed, the French healthcare system centralizes unscheduled urgent care on the ER. The aspecific respiratory symptomatology in "intermediate" patients indicates them all the more at an admission to SU or the diagnostic approach to respiratory difficulty may be carried out. It will be necessary to identify the diagnosis of the dyspneic patient and to define his virological status COVID before referring him to the appropriate units.

The investigatory propose an original strategy of dedicating entire care sectors to the care of patients admitted for dyspnea in our ER. These units will be named RECOP units.

This study would improve epidemiological knowledge of COVID-19 and ability to receive these patients within the SU.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 15 admitted to the RECOP unit for dyspnea

Exclusion Criteria:

* Patient admitted to shock for respiratory distress requiring immediate respiratory support.
* Patient under justice safeguard

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patient admitted to the RECOP unit for dyspnea will be inclued in this clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 1860 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Describe the characteristics of patients admitted to reCOP units according to their virological status vis-à-vis COVID-19 | 30 days
  The virological condition will be taken with PCR tests on naso-pharyngeal samples or on sputum for patients taking

SECONDARY OUTCOMES:
Develop a predictive model of the risk of being COVID for patients admitted to the emergency room for dyspnea | 0 days
  demographic variables, usual history and treatments, episode characteristics (symptomatology, evolution, treatment taken) and data from the initial clinical examination will be collected by doctor

OTHER OUTCOMES:
Virological status | 30 days
  Virological status will be collected by a phone call at the patient
Mortality status | 30 days
  Mortality status will be collected by a phone call at the patient

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Balen, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No